CLINICAL TRIAL: NCT05902481
Title: The Effect of Mixed Reality Technology-Based Breastfeeding Counseling on Breastfeeding Success and Self-Efficacy of Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Seda Guray, Research assistant, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 127
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breastfeeding; Breast Milk Expression; Pregnancy Related
Keywords: Breast milk; Breastfeeding; Breastfeeding counseling; Antenatal period; Mixed reality technology
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: In the study, "Block Randomization" method, which is one of the fixed probability randomization methods, will be used in order to ensure homogeneity between the groups and to eliminate selection bias. Pregnant women who meet the criteria for inclusion in the study according to block randomization will be homogeneously distributed to each training group according to their gestational week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Introductory Information Form, Antenatal Breastfeeding Self-Efficacy Scale will be applied as a pre-test after obtaining informed consent from the pregnant women who are between the 6th and 7th weeks of age.
  After the pre-test is applied, pregnant women will be given breastfeeding counseling based on mixed reality technology.
  Interventions: Other: Education
- Control Group (No Intervention): Introductory Information Form, Antenatal Breastfeeding Self-Efficacy Scale will be applied as a pre-test after obtaining informed consent from the pregnant women in the third trimester who agreed to participate in our study and met the inclusion criteria.
  After the pre-test is applied, standard breastfeeding counseling will be given to pregnant women with Power Point technique.

INTERVENTIONS:
Other: Education — education about breastfeeding with mixed reality technology.
  Arms: Intervention Group

SUMMARY:
Breast-feeding; It is the basic step of newborn, maternal and community health. Breastfeeding counseling, which is planned to encourage, initiate and continue breastfeeding in line with the recommendations of the World Health Organization, is extremely important in order to achieve the Sustainable Development Goals. Breastfeeding counseling with mixed reality technology will contribute to the literature.

The research will be carried out between January 2023 and December 2024 in the hospitals in Mersin with a delivery room. The universe will consist of all pregnant women who come to the obstetrics clinics of the specified hospitals for follow-up purposes. G Power 3.1 program was used for sampling. By using the G Power 3.1 program in the sample calculation (30); According to the Cohen Guidelines (Cohen's d); effect size was 0.5, power was 0.80, and significance level was 0.05. It was calculated as 102 people, with at least 51 people in the intervention group and at least 51 people in the control group. The sample number was determined as 112 pregnant women to receive 10% (5 each) for the intervention and control groups in case the participants dropped out of the study. In the study, "Block Randomization" method, which is one of the fixed probability randomization methods, will be used in order to ensure homogeneity between the groups and to eliminate selection bias.

In the intervention group; Introductory Information Form, Antenatal Breastfeeding Self-Efficacy Scale will be applied as a pre-test to pregnant women in their 3rd trimester and breastfeeding counseling based on mixed reality technology will be given. The LATCH Breastfeeding Diagnosis and Evaluation Scale and Postpartum Breastfeeding Self-Efficacy Scale will be filled in within 24 hours and on the 7th day after giving birth. The same steps will be performed for the pregnant women in the control group, and unlike the intervention group, counseling will be applied with Power Point technique instead of mixed reality technology. Statistical analyzes will be made using a package program called SPSS (IBM SPSS Statistics 24). In descriptive statistical analysis, mean, standard deviation, median, frequency, percentile, minimum and maximum values will be calculated. Descriptive, parametric and nonparametric statistical analysis methods will be used in the analysis of the data.

Various studies have been conducted in Turkey using different methods on breastfeeding counseling, but no study has been found in which breastfeeding counseling was provided with mixed reality technology. Therefore, a randomized controlled experimental type study will be conducted to evaluate the effect of mixed reality technology-based breastfeeding counseling on breastfeeding success and self-efficacy of women.

DETAILED DESCRIPTION:
No study has been found in Turkey that provides breastfeeding counseling with mixed reality technology. It is predicted that counseling provided with the use of mixed reality technology will increase breastfeeding self-efficacy and success. It is envisaged that the results obtained will be presented in scientific environments and used as an evidence-based practice in increasing both the rate and success of breastfeeding after being published as an article. The results of a randomized controlled trial with high evidential value are expected to be available for use by both healthcare professionals and mothers. By helping the results of the study to realize the recommendations of the World Health Organization regarding breastfeeding; It is thought that it will benefit newborn, maternal and community health, thus making a significant contribution to the promotion, initiation and maintenance of breastfeeding, which is the first step towards achieving the Sustainable Development Goals.In order to evaluate the effect of breastfeeding counseling based on mixed reality technology on breastfeeding success and self-efficacy of women, it will be conducted in a randomized controlled experimental type.

Methods The research will be carried out between January 2023 and December 2024 in the hospitals in Mersin with a delivery room.

The population of the study will be composed of pregnant women who applied to the obstetrics and gynecology outpatient clinics of hospitals with delivery rooms in Mersin between January 2023 and December 2024 for follow-up. G Power 3.1 program was used for sampling. By using the G Power 3.1 program in the sample calculation (30); According to the Cohen Guidelines (Cohen's d); effect size was 0.5, power was 0.80, and significance level was 0.05. It was calculated as a total of 102 people, with at least 51 for the intervention group (the group given breastfeeding counseling based on mixed reality technology) and at least 51 for the control group (the group where breastfeeding counseling was given with the standard education method). The sample number of the study group was determined as 112 pregnant women, 10% for the intervention group and 10% (5 people) for the control group, against the possibility of the participants dropping out of the study.

Data Collection Intervention Group Data Collection in the Prenatal Period 38-40 students who agreed to participate in our study and met the inclusion criteria. Introductory Information Form, Antenatal Breastfeeding Self-Efficacy Scale will be applied as a pre-test after obtaining informed consent from the pregnant women who are between the 6th and 7th weeks of age. The data will be collected by face-to-face interview technique and is expected to take about 15 minutes.

After the pre-test is applied, pregnant women will be given breastfeeding counseling based on mixed reality technology. Breastfeeding counseling; It is an educational program that includes breast milk and its properties, benefits of breast milk for mother and baby, breast anatomy, breastfeeding positions, expressing and storing breast milk. This counseling will be applied to pregnant women with mixed reality technology and will take approximately 20 minutes.

Data Collection in the Postpartum Period The LATCH Breastfeeding Diagnosis and Evaluation Scale will be filled by the researcher by observation within the first 24 hours after the pregnant women in the intervention group participating in our study give birth. Postpartum Breastfeeding Self-Efficacy Scale will be applied as a post-test. Data collection will take approximately 15 minutes.

The LATCH Breastfeeding Diagnosis and Evaluation Scale will be filled by the researcher through observation on the 7th day after giving birth to the pregnant women in the intervention group participating in our study. Postpartum Breastfeeding Self-Efficacy Scale will be applied as a posttest repetition. The interview will be concluded by completing the Postpartum Period Status and Satisfaction Evaluation Form. Data collection will take approximately 15 minutes.

Control Group Data Collection in the Prenatal Period Introductory Information Form, Antenatal Breastfeeding Self-Efficacy Scale will be applied as a pre-test after obtaining informed consent from the pregnant women in the third trimester who agreed to participate in our study and met the inclusion criteria. The data will be collected by face-to-face interview technique and is expected to take about 15 minutes.

After the pre-test is applied, standard breastfeeding counseling will be given to pregnant women with Power Point technique. It is an educational program that includes breastfeeding counseling, breast milk and its properties, the benefits of breast milk for mother and baby, breast anatomy, breastfeeding positions, expressing and storing breast milk. This counseling will be applied to pregnant women with Power Point technique and it will take about 20 minutes.

Data Collection in the Postpartum Period The LATCH Breastfeeding Diagnosis and Evaluation Scale will be filled by the researcher through observation within the first 24 hours after the pregnant women in the control group participating in our study give birth. Postpartum Breastfeeding Self-Efficacy Scale will be applied as a post-test. Data collection will take approximately 15 minutes.

The LATCH Breastfeeding Diagnosis and Evaluation Scale will be filled by the researcher through observation on the 7th day after giving birth to the pregnant women in the intervention group participating in our study. Postpartum Breastfeeding Self-Efficacy Scale will be applied as a posttest repetition. The interview will be concluded by completing the Postpartum Period Status and Satisfaction Evaluation Form. Data collection will take approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 38-40. Continuing pregnancy between gestational weeks,
* Primigravida,
* Those who have not received a planned breastfeeding training before,
* Pregnant women who agree to participate in the study will be included.

Exclusion Criteria:

* Having a risky pregnancy,
* Postpartum mother and/or baby have a health condition that prevents breastfeeding,
* Having multiple pregnancy,
* The mother and/or baby hospitalized for the first 7 days,
* Can't speak or understand Turkish,
* Women with intellectual disability and serious mental disorders will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Antenatal Breastfeeding Self-Efficacy Scale | 1 day
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed.This scale assesses how competent mothers feel about breastfeeding.The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy. This scale can be applied both in the antenatal and postnatal periods.
Postpartum Breastfeeding Self-Efficacy Scale | 1 day
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed.This scale assesses how competent mothers feel about breastfeeding.The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy. This scale can be applied both in the antenatal and postnatal periods.The difference of the antenatal form of the scale from the postnatal form is the use of the phrase "future tense" in the scale items.
LATCH Breastfeeding Diagnosis and Evaluation Scale | 1 day
  The LATCH Breastfeeding Diagnostic and Evaluation Scale was developed by Jensen et al. in 1994 (36). The Turkish validity and reliability of the scale were performed by Demirhan and Pek in 1997, Koyun in 2001, and Yenal and Okumuş in 2003 (37,38). The LATCH Breastfeeding Diagnostic and Evaluation Scale is a scale filled by the researcher through observation.
Postpartum Breastfeeding Self-Efficacy Scale | 1 day
  It was developed by the researcher in line with the literature in order to determine the characteristics of infants and breastfeeding in the postnatal period. In the form, data related to the birth process such as the week of gestation, the mode of delivery and the situation of experiencing problems during delivery; There are 11 questions questioning the breastfeeding experience, such as the baby's gender, height and weight, the time of first breastfeeding, problems during breastfeeding, and the first food given to the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, Study Director — Cukurova University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Alliance for Breastfeeding Action (WABA). Messages for World Health Day 2022 - Breastfeeding Is A Climate-smart Decision. https://waba.org.my/ . Erişim Tarihi: 12.10.2022
- [Background] Chowdhury R, Sinha B, Sankar MJ, Taneja S, Bhandari N, Rollins N, Bahl R, Martines J. Breastfeeding and maternal health outcomes: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):96-113. doi: 10.1111/apa.13102. PMID 26172878
- [Background] Krol KM, Grossmann T. Psychological effects of breastfeeding on children and mothers. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2018 Aug;61(8):977-985. doi: 10.1007/s00103-018-2769-0. PMID 29934681
- [Background] Tewabe T. Prelacteal Feeding Practices among Mothers in Motta Town, Northwest Ethiopia: A Cross-sectional Study. Ethiop J Health Sci. 2018 Jul;28(4):393-402. doi: 10.4314/ejhs.v28i4.5. PMID 30607052
- [Background] Rozga MR, Kerver JM, Olson BH. Self-reported reasons for breastfeeding cessation among low-income women enrolled in a peer counseling breastfeeding support program. J Hum Lact. 2015 Feb;31(1):129-37; quiz 189-90. doi: 10.1177/0890334414548070. Epub 2014 Aug 26. PMID 25158829
- [Background] Martin-Iglesias S, Santamaria-Martin MJ, Alonso-Alvarez A, Rico-Blazquez M, Del Cura-Gonzalez I, Rodriguez-Barrientosn R, Barbera-Martin A, Sanz-Cuesta T, Isabel Coghen-Vigueras M, de Antonio-Ramirez I, Durand-Rincon I, Garrido-Rodriguez F, Geijo-Rincon MJ, Mielgo-Salvador R, Morales-Montalva MS, Reviriego-Gutierrez MA, Rivero-Garrido C, Ruiz-Calabria M, Santamaria-Mechano MP, Santiago-Fernandez R, Sillero-Quintana MI, Soto-Almendro B, Terol-Claramonte M, Villa-Arranz M. Effectiveness of an educational group intervention in primary healthcare for continued exclusive breast-feeding: PROLACT study. BMC Pregnancy Childbirth. 2018 Feb 26;18(1):59. doi: 10.1186/s12884-018-1679-3. PMID 29482516
- [Background] Alakaam A. Demand for Lactation Leads to Flowing Supply of Success: Support Requested from States to Improve Breastfeeding Practices. J Midwifery Womens Health. 2019 Nov;64(6):699-702. doi: 10.1111/jmwh.12977. Epub 2019 Jul 9. No abstract available. PMID 31287205
- [Background] Nicholson WK, Beckham AJ, Hatley K, Diamond M, Johnson LS, Green SL, Tate D. The Gestational Diabetes Management System (GooDMomS): development, feasibility and lessons learned from a patient-informed, web-based pregnancy and postpartum lifestyle intervention. BMC Pregnancy Childbirth. 2016 Sep 21;16(1):277. doi: 10.1186/s12884-016-1064-z. PMID 27654119
- [Background] Khorshidifard M, Amini M, Dehghani Mr, Zaree N, Pishva N & Zarifsanaiey N. Assessment of breastfeeding education by face to face and small-group education methods in mothers' self-efficacy in Kazeroun Health Centers in 2015. Women's Health Bulletin, 2017, 4(3):2-6.